CLINICAL TRIAL: NCT00000971
Title: A Phase I/II Dose-Ranging, Pharmacokinetic, Drug Interaction, Safety and Preliminary Efficacy Study of Oral Clarithromycin Granules for Suspension, in Combination With Zidovudine or Dideoxyinosine, in the Treatment of Disseminated Mycobacterium Avium Complex Infections in Pediatric Patients With AIDS
Brief Title: The Safety and Effectiveness of Clarithromycin Plus Zidovudine or Dideoxyinosine in the Treatment of Mycobacterium Avium Complex (MAC) Infections in Children With AIDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 178; NCI 91 C-53
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 1996-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Didanosine; Drug Evaluation; Drug Interactions; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Clarithromycin; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Clarithromycin
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To evaluate three doses of clarithromycin in children with AIDS and Mycobacterium avium complex (MAC) infection who are receiving concurrent antiretroviral therapy.

Before more extensive evaluation of this promising drug for treatment of MAC infection in children can be done, it is important to study the pharmacokinetics of this drug in this population, to get information regarding its use in pediatric patients receiving currently available antiretroviral drugs, and to get information on the antimycobacterial activity of this drug.

DETAILED DESCRIPTION:
Before more extensive evaluation of this promising drug for treatment of MAC infection in children can be done, it is important to study the pharmacokinetics of this drug in this population, to get information regarding its use in pediatric patients receiving currently available antiretroviral drugs, and to get information on the antimycobacterial activity of this drug.

Patients that are included are HIV infected and have started zidovudine (AZT) or didanosine (ddI) at least 4 weeks before entry into this study. Patients continue taking the medications at prescribed doses. In addition they also take clarithromycin. Patients continue treatment with AZT or ddI plus clarithromycin for 12 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis treatment for Pneumocystis carinii pneumonia.
* Topical antivirals.

Prior Medication: Required:

* Zidovudine (AZT), 90 - 180 mg/m2 q6h, or didanosine (ddI), 60 - 120 mg/m2 q8h for 4 weeks prior to study entry.

Patients must have the following:

* Diagnosis of AIDS and Mycobacterium avium complex.
* Ability to tolerate therapy with zidovudine or didanosine at specified dosages.
* Written consent from a parent or legal guardian.
* Willing to comply with all procedures and scheduled visits. Relatively stable clinical condition.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of significant depressive disorder.
* History of allergy to macrolide antibiotics.
* Presence of acute bacterial infection or acute onset of opportunistic infection as listed in protocol.

Patients with the following are excluded:

* Presence of current opportunistic infection other than Mycobacterium avium complex defined as systemic candidemia, cryptosporidiosis, isosporiasis, toxoplasmosis, pneumocystosis, salmonellosis, or acute bacterial infection.

Prior Medication:

Excluded within 30 days of study entry:

* Systemic antimycobacterial drugs, myelosuppressive drugs, nephrotoxic agents, cytotoxic or experimental chemotherapy, or antiviral drugs.

Active alcohol or drug use sufficient in the opinion of the investigator to prevent adequate compliance with medication regimen and clinic visits.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Overall Officials: Pizzo P, Study Chair; Husson R, Study Chair
Locations (2):
- United States (2):
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Natl Cancer Institute / HIV / AIDS Malignancy Branch, Bethesda, Maryland

REFERENCES:
- [Background] Husson RN, Ross LA, Sandelli S, Inderlied CB, Venzon D, Lewis LL, Woods L, Conville PS, Witebsky FG, Pizzo PA. Orally administered clarithromycin for the treatment of systemic Mycobacterium avium complex infection in children with acquired immunodeficiency syndrome. J Pediatr. 1994 May;124(5 Pt 1):807-14. doi: 10.1016/s0022-3476(05)81380-0. PMID 8176574